CLINICAL TRIAL: NCT02270710
Title: Immune Deregulation in Patients With SLE
Brief Title: Molecular Mechanisms Characteristics in Systemic Lupus Erythematous Autoimmune Disease
Acronym: SLE
Status: Withdrawn | Type: Observational
Why Stopped: Research direction changed
Sponsor: Weill Medical College of Cornell University (Other)
Collaborators: Hospital for Special Surgery, New York (Other)
Responsible Party: Sponsor
Other Study IDs: 1311014560
Record Dates: First submitted 2014-10-16; First posted 2014-10-21 (Estimated); Last update posted 2017-05-24 (Actual); Status verified 2017-05

CONDITIONS: Systemic Lupus Erythematosus
MeSH Terms: conditions — Lupus Erythematosus, Systemic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — Blood
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Healthy Subjects: Overall in good health Provide informed consent Male and females, age 18 years and older Nonsmokers
- SLE Subjects: Enrolled by Hospital for Special Surgery Diagnosed with Systemic Lupus Erythematosus

SUMMARY:
It is well known that the deregulation of immune responses plays a major role in many autoimmune diseases, such as Systemic Lupus Erythematosus (SLE). The main objective of this protocol is to determine whether the expression and/or function of specific molecules are deregulated in the immune cells of patients with SLE. By examining IRF4, IRF5, IBP/Def6, SWAP-70, Rock1, Rock2, and specific signaling molecules involved in the responsiveness to sex hormones, the investigators hypothesize that the deregulation in the expression and function of these molecules will result in abnormalities in the functioning of the immune cells, which is a key factor in autoimmunity.

Peripheral blood lymphocytes from healthy controls and patients with SLE will be collected and compared in order to determine if specific immune cells (IL-17 and IL-21) are deregulated in patients with SLE and if this deregulation affects their functioning. Specifically, immune cells will be isolated from the blood and then subject to scientific testing (QPCR, Western blotting, immunofluorescence assays, ELISA and FACS analysis) to see if the expression and function of these cells is related to the mechanism behind SLE. This will be a case control study, where cases of SLE will be compared to controls of healthy volunteers to assess risk factors. As these healthy volunteers are providing samples solely for research purposes, there is no standard of care for these volunteers, with the exception of a positive HIV result during screening. The Department of Genetic Medicine will enroll healthy controls and the Hospital for Special Surgery will enroll subjects with Systemic Lupus Erythematosus (SLE) for a comparative analysis of the two cohorts. Laboratory testing on all blood samples will be done at the Hospital for Special Surgery.

DETAILED DESCRIPTION:
This will be a case control study, where cases of SLE will be compared to controls of healthy volunteers to assess risk factors. As these healthy volunteers are providing samples solely for research purposes, there is no standard of care for these volunteers, with the exception of a positive HIV result during screening. The Department of Genetic Medicine will enroll healthy controls and the Hospital for Special Surgery will enroll subjects with Systemic Lupus Erythematosus (SLE) for a comparative analysis of the two cohorts (Table I). Laboratory testing on all blood samples will be done at the Hospital for Special Surgery.

Table I. Site Recruitment1

WCMC Healthy Subjects 20 HSS Subjects with SLE 20 Total 40

ELIGIBILITY:
Inclusion Criteria:

* Must provide informed consent
* Males and females, age 18 years and older
* Healthy Nonsmokers

Exclusion Criteria:

If the subject has

* Rheumatic disease
* Diabetes
* SLE or lupus
* Autoimmune disease
* Active infection or pregnancy
* HIV infection

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy Subjects
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2013-04; Primary Completion 2016-10 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
Determine the molecules that play a role in onset of SLE and autoimmune disease | 1 year
  Immune cells isolated from blood samples of healthy and SLE subjects IRF4, IRF5, IBP/Def6, SWAP-70, Rock1, Rock2 molecules expression examined through scientific testing (QPCR, Western blotting, immunofluorescence assays, ELISA and FACS analysis)

CONTACTS AND LOCATIONS:
Overall Officials: Ronald G Crystal, MD, Principal Investigator — Department of Genetic Medicine
Locations (1):
- Weill Medical College of Cornell University, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided